CLINICAL TRIAL: NCT00217087
Title: Endoscopic Therapy of Early Cancer in Barretts Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kenneth K. Wang, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1399-05; R01CA111603 (NIH)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2015-09-25 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Early Stage Esophageal Adenocarcinoma; Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopic Mucosal Resection; Photochemotherapy; Dihematoporphyrin Ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic Mucosal Resection (Other): Patients will undergo endoscopic mucosal resection at time of endoscopy if indicated.
  Interventions: Procedure: Endoscopic Mucosal Resection
- Photodynamic Therapy (Other): Patients will have endoscopic mucosal resection with photodynamic therapy.
  Interventions: Procedure: Endoscopic Mucosal Resection; Procedure: Photodynamic Therapy

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection — Endoscopic mucosal resection at time of endoscopy if indicated.
Procedure: Photodynamic Therapy — Porfimer sodium 2mg/kg
  Other Names: Photofrin
  Arms: Photodynamic Therapy

SUMMARY:
This study is being done to see if treatment for esophageal cancer can be done using endoscopy for patients ineligible for surgical or radiological therapy. The standard method of treating this type of cancer is surgical removal of the esophagus. The study will determine if removing just the cancer with endoscopy is enough treatment or if the addition of another treatment called photodynamic therapy (treatment with a red light and a drug called sodium porfimer) is needed.

DETAILED DESCRIPTION:
Participant visit requirements: Screening visit which will last 1 - 2 days, if assigned to photodynamic therapy, there will be a 3 day visit for treatment. Participants must return for a 1 day visit every three months for one year.

ELIGIBILITY:
Inclusion Criteria:

* Non-recurrent adenocarcinoma in Barrett's Esophagus confirmed by two experienced gastrointestinal pathologists
* No evidence of submucosal invasion
* No evidence of metastatic disease in either regional or distal lymph nodes, or other organs
* Pre-entry CT scans of the upper abdomen and chest and Endoscopic Ultrasound (EUS) of the tumor and regional lymph nodes are required. Fusion PET scans are suggested for any indeterminate lesions
* Zubrod Performance Status 0-1
* Participants must be have oral intake of greater than 1700 calories a day
* Patient must not have had a second malignancy, other than curable non-melanoma skin cancer or cervical cancer in situ, unless disease free for greater than or equal to 3 years and deemed cured by their hematologist and/or oncologist
* Staging procedures should be performed prior to study entry
* All patients or legally authorized representative must sign a study-specific informed consent prior to randomization.

Exclusion criteria:

* Prior major esophageal surgery
* Patients who are unable to tolerate endoscopic procedures
* Due to the possible toxic effects of photodynamic therapy and endoscopic sedation to embryos, pregnant or lactating women or men unable or unwilling to practice contraception are excluded
* Patients with an uncontrolled diabetes, heart disease, or hypertension
* Patient and/or legally authorized representative who are unable to comprehend the study requirements or who are not likely to comply with the study parameters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2005-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K. Wang, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from December 1, 2005 thru April 26, 2011 at Mayo Clinic in Rochester, Minnesota.
Pre-assignment Details: We intended to recruit 100 patients with early cancer and were able to recruit a total of 124 patients in this single center randomized trial. A total of 73 patients could actually be randomized due to inability to completely remove the cancer, finding evidence of high risk of metastasis, or refusing randomization to photodynamic therapy.
Groups:
- Photodynamic Therapy: Patients will have endoscopic mucosal resection (if indicated at time of endoscopy) followed by photodynamic therapy.
Period: Overall Study
Arm/Group | Endoscopic Mucosal Resection | Photodynamic Therapy
Started | 36 | 37
Completed | 25 | 17
Not Completed | 11 | 20
Not completed — decided to have esophagectomy | 1 | 2
Not completed — completed less than 12 months return | 10 | 18

BASELINE CHARACTERISTICS:
Groups:
- Endoscopic Mucosl Resection: patients will undergo endoscopic mucosal resection at time of endoscopy if indicated
- Total: Total of all reporting groups
Arm/Group | Endoscopic Mucosl Resection | Photodynamic Therapy | Total
Number analyzed (Participants) | 36 | 37 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 23 | 25 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 33 | 31 | 64
Region of Enrollment [Number; unit: participants]
  United States | 36 | 37 | 73

OUTCOME MEASURES:

1. Primary Outcome: Level of Dysplasia on Histology at 12 Months
Description: All specimens were reviewed by two expert GI pathologists for presence of and/or level of dysplasia in Barrett's Esophagus
Time Frame: 12 months post therapy
Population: 4 participants in the photodynamic therapy group completed at least 3 but less than 12 months follow up post therapy, so they were not included in this analysis.
Measure: Number; unit: paricipants
Arm/Group | Endoscopic Mucosal Resection | Photodynamic Therapy
Number analyzed (Participants) | 25 | 13
paricipants
  Decreases in dysplasia from enrollment | 10 | 11
  No improvement or worsened level of dysplasia | 15 | 2
Statistical Analysis 1: Comparison: Endoscopic Mucosal Resection vs Photodynamic Therapy; Test type: Superiority or Other; p = 0.0098, Fisher Exact

2. Primary Outcome: Fluorescence In Situ Hybridization (FISH) Markers at 12 Months.
Description: Whether or not positive fish markers measured by polysomy were associated with outcomes.
  Markers in this study include: 9q21 /017q (her2) / 8q24/ 20q / CEP17 / 17p. Polysomy and Trisomy were documented.
Time Frame: 12 months post therapy
Population: 4 participants in the PDT group completed at least 3 months of follow up but not 12 months
Measure: Number; unit: participants
Groups:
- Endoscopic Mucosal Resection FISH Polysomy Negative; Photodynamic Therapy FISH NEGATIVE: FISH cytology results prior to therapy were negative
- Endoscopic Mucosal Resection FISH Positive Positive; Photodynamic Therapy FISH POSITIVE: FISH cytology results were positive prior to therapy
Arm/Group | Endoscopic Mucosal Resection FISH Polysomy Negative | Endoscopic Mucosal Resection FISH Positive Positive | Photodynamic Therapy FISH POSITIVE | Photodynamic Therapy FISH NEGATIVE
Number analyzed (Participants) | 11 | 13 | 8 | 5
participants
  Decrease level of dysplasia post therapy | 7 | 8 | 6 | 5
  no change or worsening of dysplasia post therapy | 4 | 5 | 2 | 0
Statistical Analysis 1: Comparison: Endoscopic Mucosal Resection FISH Polysomy Negative vs Endoscopic Mucosal Resection FISH Positive Positive; Test type: Superiority or Other; p = 0.34, Chi-squared

3. Primary Outcome: Change in Quality of Life
Description: Quality of life in both groups (EMR and EMR with photodynamic therapy) SF36
Time Frame: end of study
Population: 25 patients did not return completed SF36 at 12 month of follow up their results were not used in final analysis.
Measure: Number; unit: participants
Groups:
- Endoscopic Mucosal Resection: Patients will undergo EMR at time of endoscopy if indicated.
- Endoscopic Mucosal Resection and Photodynamic Therapy: Patients will have EMR (if indicated at time of endoscopy) followed by photodynamic therapy
Arm/Group | Endoscopic Mucosal Resection | Endoscopic Mucosal Resection and Photodynamic Therapy
Number analyzed (Participants) | 10 | 6
participants
  qaulity of life remained the same of improved | 9 | 6
  decrease in qualify of life | 1 | 0
Statistical Analysis 1: Comparison: Endoscopic Mucosal Resection vs Endoscopic Mucosal Resection and Photodynamic Therapy; Test type: Superiority or Other; p = 0.2, Chi-squared; the only participant who reported a decrease quality of life related that to a recent surgery not their esophagus

ADVERSE EVENTS:
Time Frame: 6 years, 2 months
Arm/Group | Endoscopic Mucosl Resection | Photodynamic Therapy
Serious Adverse Events (participants affected / at risk) | 1/36 | 4/37
Other Adverse Events (participants affected / at risk) | 3/36 | 21/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endoscopic Mucosl Resection (N=36) | Photodynamic Therapy (N=37)
Renal failure - Sepsis (Renal and urinary disorders) | 0 (0) | 1 (1) — unrelated to study participation
Respitory Failure / Sepsis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — unrelated to study participation
heart attack resulting in death (Cardiac disorders) | 1 (1) | 2 (2) — not related to study participation
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Endoscopic Mucosl Resection (N=36) | Photodynamic Therapy (N=37)
Bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) — known/anticipated risk - post endoscopic mucosal resection - treated endoscopically or observation only
Dehydration (General disorders) | 1 (1) | 1 (1) — required hospitalization with IV fluids both incidents were unrelated to study participation
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (12) — known and anticipated risk of Photodynamic therapy (Photofrin)
Atrial fibrilation (Cardiac disorders) | 1 (1) | 0 (0) — not related to study participation
Pain (Gastrointestinal disorders) | 0/0 (0) | 1 (1) — Participant had pain last longer than is anticipated after photodynamic therapy, treated with medication
Dysphagia (Gastrointestinal disorders) | 0 (0) | 6 (6) — known and anticipated event post photodynamic therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No